CLINICAL TRIAL: NCT07148635
Title: Electrical Dry Needling Versus Sham Dry Needling in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ammar Sanaullah, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0026
Record Dates: First submitted 2025-08-23; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: Electrical Dry Needling; Myofascial Trigger Points; Myofascial Pain Syndrome; Kinesiophobia; Sham Dry Needling
MeSH Terms: conditions — Myofascial Pain Syndromes; Kinesiophobia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electrical Dry Needling with Conventional Therapy (Experimental): Participants will receive electrical dry needling (EDN) applied to active myofascial trigger points in lumbar muscles (quadratus lumborum, multifidus, iliocostalis lumborum) once weekly for six weeks. Fine monofilament needles will be inserted into trigger points and connected to a low-frequency electrical stimulator (2-10 Hz) for 10-15 minutes per session. In addition, participants will follow a standardized physiotherapy program including core strengthening, lumbar and hamstring stretching, posture education, and a home-based exercise plan.
  Interventions: Procedure: Electrical Dry Needling (EDN)
- Sham Dry Needling with Conventional Therapy (Placebo Comparator): Participants will receive sham dry needling (SDN) once weekly for six weeks. Needles will be applied superficially or with blunt instruments at the same anatomical points as the experimental arm, but without penetration into muscle tissue and without electrical stimulation. Alongside SDN, participants will receive the same standardized physiotherapy program as the experimental group, including core strengthening, stretching, posture education, and a home-based exercise plan.
  Interventions: Procedure: Sham Dry Needling (SDN)

INTERVENTIONS:
Procedure: Electrical Dry Needling (EDN) — Electrical dry needling will be performed at active myofascial trigger points in lumbar muscles (quadratus lumborum, multifidus, iliocostalis lumborum). Fine monofilament needles are inserted into trigger points and connected to a low-frequency stimulator (2-10 Hz) for 10-15 minutes per session. Treatment is delivered once weekly for six weeks by a trained physiotherapist. Participants will also receive standardized conventional physiotherapy including core strengthening, stretching, posture education, and a home-based exercise program.
  Arms: Electrical Dry Needling with Conventional Therapy
Procedure: Sham Dry Needling (SDN) — Sham dry needling will be administered at the same anatomical sites as the experimental group, using superficial or blunt needle placement without penetration into muscle tissue and without electrical stimulation. Sessions are delivered once weekly for six weeks by a trained physiotherapist. Participants will also receive the same standardized conventional physiotherapy including core strengthening, stretching, posture education, and a home-based exercise program to maintain consistency with the experimental arm.
  Arms: Sham Dry Needling with Conventional Therapy

SUMMARY:
This study will evaluate the effectiveness of electrical dry needling (EDN) compared to sham dry needling (SDN) in patients with chronic low back pain (CLBP). CLBP is a common musculoskeletal condition associated with persistent pain, functional limitations, and reduced quality of life. Myofascial trigger points (MTrPs) are often implicated in CLBP and represent a key therapeutic target.

Dry needling is a minimally invasive procedure where fine needles are inserted into trigger points to release muscle tension and alleviate pain. Electrical dry needling is an advanced variation that applies low-frequency electrical stimulation through the inserted needles, potentially enhancing therapeutic effects. However, evidence is limited regarding its superiority over sham procedures.

In this randomized controlled trial, 70 adult participants with CLBP persisting for at least three months will be randomly assigned to one of two groups:

Group A (EDN + Conventional Therapy): Patients will receive electrical dry needling at active MTrPs combined with a structured physiotherapy program.

Group B (SDN + Conventional Therapy): Patients will receive sham dry needling at the same anatomical sites (using superficial or blunt needle placement without penetration) alongside the same physiotherapy program.

Interventions will be delivered weekly for six weeks. Assessments will occur at baseline, third week, and sixth week.

Primary outcomes include:

Pain intensity (Visual Analogue Scale, VAS)

Functional disability (Roland-Morris Disability Questionnaire, RMDQ)

Kinesiophobia (Tampa Scale of Kinesiophobia, TSK)

This trial is designed to clarify the clinical value of EDN beyond placebo effects, providing evidence to guide management of CLBP.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) affects approximately 7-8% of the global population and remains a leading cause of disability and healthcare burden. Conventional management strategies, including medication, manual therapy, and exercise, often provide partial or temporary relief. Myofascial trigger points (MTrPs) are highly prevalent in CLBP and contribute to persistent pain and movement restrictions.

Dry needling has emerged as a widely used intervention to deactivate MTrPs. The technique produces a local twitch response, improves blood flow, and reduces muscle tightness. Electrical dry needling (EDN) enhances this effect by delivering low-frequency electrical stimulation through the inserted needles, which may result in improved neuromuscular relaxation and pain modulation.

Despite encouraging findings from prior studies, the literature lacks rigorous trials comparing EDN with sham dry needling (SDN) controls. Sham procedures are critical to distinguish specific treatment effects from placebo or expectancy effects. This study aims to fill that gap.

Study Design:

Randomized controlled trial (parallel groups, single-blind).

Sample size: 70 patients (35 per group), aged 18-25 years, with CLBP >3 months and confirmed active MTrPs.

Recruitment site: Social Security Hospital, Kot Lakhpat, Lahore.

Duration: 9 months after approval.

Randomization: Lottery method.

Blinding: Single-blind (assessor unaware of treatment allocation).

Interventions:

Group A (EDN + Conventional Therapy): Weekly 30-45 min sessions for 6 weeks. EDN applied at quadratus lumborum, multifidus, and iliocostalis lumborum trigger points, with low-frequency electrical stimulation (2-10 Hz, 10-15 minutes). Physiotherapy includes core strengthening, stretching, posture education, and home-based exercises.

Group B (SDN + Conventional Therapy): Same physiotherapy protocol. Sham needling applied with superficial or blunt needles without tissue penetration; no electrical stimulation.

Outcome Measures:

Pain intensity (VAS)

Functional disability (Roland-Morris Disability Questionnaire)

Kinesiophobia (Tampa Scale of Kinesiophobia)

Data Collection: Baseline, 3rd week, and 6th week.

Statistical Analysis: Data will be analyzed using SPSS v24. Descriptive statistics will summarize demographics. Normality will be tested (Shapiro-Wilk/Kolmogorov-Smirnov). Between- and within-group comparisons will be conducted using ANOVA for parametric data, or Mann-Whitney/Wilcoxon tests for non-parametric data. Significance level set at p < 0.05.

Ethical Considerations:

The study has received Institutional Research Ethics Board (IREB) approval from the University of Lahore. Informed consent will be obtained from all participants. Confidentiality, anonymity, and voluntary participation will be ensured. Participants may withdraw at any time without penalty.

Potential Impact:

This study will provide high-quality evidence on the clinical effectiveness of EDN compared to SDN in CLBP patients. If successful, EDN may be integrated into physiotherapy practice as an evidence-based intervention for reducing pain, disability, and fear of movement in this population.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female gender will be included (Fernández-Carnero, 2021).
* Clinically diagnosed of chronic low back pain persisting for at least three months (Tüzün et al., 2017)
* Identifiable active myofascial trigger points in the lower back muscles, confirmed through palpation or another standardized method (Donohoe, 2016).
* Moderate to severe pain intensity, measured by a visual analog scale (VAS) (Tüzün et al., 2017)
* Sufficient cognitive and physical ability to engage in assessments and interventions (Tüzün et al., 2017)

Exclusion Criteria:

* Known hypersensitivity to needles, history of severe bleeding disorders, or any condition that contraindicates dry needling (Tüzün et al., 2017)
* Use of other physical therapy interventions or dry needling treatments in the last three months for low back pain (Fernández-Carnero, 2021).
* Presence of specific spinal conditions (e.g., disc herniation, spinal stenosis, fractures, or recent spinal surgeries) (Tüzün et al., 2017)
* History of neurological conditions affecting movement, sensation, or pain perception, such as multiple sclerosis or peripheral neuropathy (Donohoe, 2016)
* Pregnant women will be excluded due to potential risks associated with the interventions (Tüzün et al., 2017)
* Unstable psychiatric conditions or active substance abuse that could interfere with participation or adherence to study procedures

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2025-04-09 (Actual); Primary Completion 2025-08-11 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (Visual Analogue Scale, VAS) | Baseline, 3rd week, and 6th week
  Pain will be assessed using a 10-cm Visual Analogue Scale, where 0 indicates "no pain" and 10 indicates "worst imaginable pain." This provides a validated, subjective measure of current pain intensity.
Functional Disability (Roland-Morris Disability Questionnaire, RMDQ) | Baseline, 3rd week, and 6th week
  Functional disability will be evaluated using the 24-item Roland-Morris Disability Questionnaire. Scores range from 0 to 24, with higher scores indicating greater disability and functional limitations due to low back pain.
Kinesiophobia (Tampa Scale of Kinesiophobia, TSK) | Baseline, 3rd week, and 6th week
  Fear of movement will be measured using the 17-item Tampa Scale of Kinesiophobia (TSK). Items are scored on a 4-point Likert scale (range 17-68), with higher scores indicating greater fear of movement and injury.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tuzun EH, Gildir S, Angin E, Tecer BH, Dana KO, Malkoc M. Effectiveness of dry needling versus a classical physiotherapy program in patients with chronic low-back pain: a single-blind, randomized, controlled trial. J Phys Ther Sci. 2017 Sep;29(9):1502-1509. doi: 10.1589/jpts.29.1502. Epub 2017 Sep 15. PMID 28931976